CLINICAL TRIAL: NCT01513070
Title: A Randomized Double-blind Placebo-controlled Clinical Trials of the Blood-quickening Stasis-transforming Formula Quick-Acting Heart Reliever for Patients With Moderate Coronary Stenosis
Brief Title: A Clinical Trials of Quick-Acting Heart Reliever for Moderate Coronary Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, President of Guang'anmen Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUXIAOJIUXIN2010
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Stenosis; Coronary Heart Disease
Keywords: Quick-Acting Heart Reliever; Coronary Artery Stenosis; Coronary Heart Disease; Suxiao Jiuxin Pill; Chinese Herbal Drugs; Traditional Chinese Medicine; Chinese Medicine; Angina Pectoris; Isosorbide Dinitrate; Myocardial Perfusion Imaging; Clinical Trial
MeSH Terms: conditions — Coronary Stenosis; Coronary Disease; Angina Pectoris | interventions — Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quick-Acting Heart Reliever group (Experimental): Drug: Quick-Acting Heart Reliever and Placebo of isosorbide dinitrate and Aspirin Enteric-coated Tablets
  Interventions: Drug: Quick-Acting Heart Reliever; Drug: Placebo of Isosorbide Dinitrate; Drug: Aspirin Enteric-coated Tablets
- Isosorbide Dinitrate group (Active Comparator): Isosorbide Dinitrate and Placebo of Quick-Acting Heart Reliever and Aspirin Enteric-coated Tablets
  Interventions: Drug: Isosorbide Dinitrate; Drug: Placebo of Quick-Acting Heart Reliever; Drug: Aspirin Enteric-coated Tablets

INTERVENTIONS:
Drug: Quick-Acting Heart Reliever — Quick-Acting Heart Reliever，200mg，tid，po. for six months
  Other Names: Suxiao Jiuxin Pill
  Arms: Quick-Acting Heart Reliever group
Drug: Isosorbide Dinitrate — Isosorbide Dinitrate，10mg，tid，po. for six months
  Other Names: Cedocard，Nitrosorbide， Vascardin
  Arms: Isosorbide Dinitrate group
Drug: Placebo of Isosorbide Dinitrate — Placebo of Isosorbide Dinitrate，10mg，tid，po. for six months
  Arms: Quick-Acting Heart Reliever group
Drug: Aspirin Enteric-coated Tablets — Aspirin Enteric-coated Tablets，100mg，qd，po. for six months
  Arms: Quick-Acting Heart Reliever group
Drug: Placebo of Quick-Acting Heart Reliever — Placebo of Quick-Acting Heart Reliever，200mg，tid，po. for six months
  Arms: Isosorbide Dinitrate group
Drug: Aspirin Enteric-coated Tablets — Aspirin Enteric-coated Tablets，100mg，qd，po. for six months
  Arms: Isosorbide Dinitrate group

SUMMARY:
This study investigates the effective power of angina pectoris after Quick-Acting Heart Reliever and isosorbide dinitrate interventing respectively the patients with moderate coronary stenosis for six months. At the same time, the studying will assess the plaque, myocardial blood-supplying,quality of life and observe the end point of the heart (including the myocardial revascularization, death and myocardial infarction). The purpose is to study the function of the blood-quickening stasis-transforming formula Quick-Acting Heart Reliever for moderate coronary stenosis lesions.

DETAILED DESCRIPTION:
Blood-quickening stasis-transforming medicinal of Chinese medicinal can ameliorate clinical symptoms of coronary artery disease. Quick-Acting Heart Reliever is one of blood-quickening stasis-transforming medicinals to relieve angina pectoris in clinic and is especially benefit for the patients with moderate coronary stenosis who need not coronary revascularization only have medical treatment. But there is no randomized evidence that established the beneficial effects of blood-quickening stasis-transforming medicinals to treat moderate coronary stenosis lesions. This study is a randomized double-blind placebo-controlled clinical trials. A total of 120 consecutive participants with at least one moderate coronary stenosis lesion (diameter stenosis 50-75%) will be randomized to two groups: group 1(n =60) will receive Quick-Acting Heart and the placebo of isosorbide dinitrate, patients in group 2(n = 60) will receive isosorbide dinitrate and the placebo of Quick-Acting Heart for six months. The myocardial perfusion imaging and the coronary CT angiography will be used to evaluate the effective power of angina pectoris,myocardial blood-supplying，the quality and volume of the plaque, diameter stenosis after treating after 6 months and the end point of the heart (including death，myocardial infarction and myocardial revascularization which includes intracoronary stenting and coronary artery bypass grafting,) after 12 months. The purpose is to study the function of Quick-Acting Heart Reliever delaying percutaneous coronary intervention(PCI) for moderate coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 30-75 years of age
* Angina or CAD patient
* Diameter stenosis 50-75% in at least one main coronary artery (Confirmed by coronary arteriography or coronary CT angiography)
* Not received percutaneous coronary intervention(PCI)
* Heart blood stasis obstruction syndrome according to TCM syndrome differentiation
* Provide written informed consent.

Exclusion Criteria:

* Heart transplant or history of CABG or history of percutaneous transluminal coronary angioplasty (PTCA) with a drug-eluting stent.
* Left ventricular ejection fraction < 35%
* Acute myocardial infarction within 4 weeks prior to inclusion
* The contractive pressure > 160 mmHg or diastolic pressure >100 mmHg
* Severe valvular heart disease
* Insulin-dependent diabetes mellitus
* Serious heart, lung, liver, kidney and brain or other primary complications
* Mental patients
* Diagnosed or suspected tumor
* Allergic persons
* Pregnant, breastfeeding, or intends to become pregnant during the course of the study (females only)
* Patients not willing to or not able to give the informed consent to participate in the study
* The patients who are attending other clinical trial
* The person maybe loss for some reason such as work or life condition according to the investigator's judgement

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the effective power of angina pectoris | 6 months
  the effective power of angina pectoris after Quick-Acting Heart Reliever and isosorbide dinitrate interventing respectively the patients with morderate coronary stenosis for six months

SECONDARY OUTCOMES:
plaque | 6 months
  Assess the plaque by the coronary CT angiography
myocardium blood-supply | 6 months
  Evaluate the myocardium blood-supply by the myocardial perfusion imaging
the end point of the heart(a composite of cardiovascular events including death, nonfatal myocardial infarction,coronary revascularization, hospitalized unstable angina) | 12 months
symptoms score | 6 months
quality of life | 6 months
MMP-9 | 6 months
SCD40L | 6 months
VEGF | 6 months
bFGF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China